CLINICAL TRIAL: NCT06079450
Title: Effect of Artıfıcıal Intellıgence Based Mobıle Vırtual Assıstant Developed For Indıvıduals Wıth Dıabetes On Cost Effıcıency, Hospıtal Admıssıon Rate, Self-Care And Hypoglycemıa
Brief Title: Effect of Artıfıcıal Intellıgence Based Mobıle Vırtual Assıstant
Acronym: AI
Status: Completed | Type: Observational
Sponsor: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Gökşen POLAT, Lecturer of Internal Medicine Nursing, Izmir Tinaztepe University
Other Study IDs: IKCU
Record Dates: First submitted 2023-08-10; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diabetes
Keywords: Diabetes; mobile application; artificial intelligence; self-care; hospitalization; cost
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Artificial intelligence-based mobile application initiative was implemented for diabetes patients
  Interventions: Other: artificial intelligence based mobile application
- control group: no intervention was applied

INTERVENTIONS:
Other: artificial intelligence based mobile application — Artificial intelligence-based mobile application developed by me that includes diabetes education for individuals with diabetes.
  Groups: experimental group

SUMMARY:
Aim: This study was conducted experimentally to examine the effect of artificial intelligence-based mobile virtual assistant developed for individuals with diabetes on cost, hospitalization rate, self-care and hypoglycemia.

Methods: The research is multi-stage and designed as three stages in itself. According to this; development of the mobile application in the first and second stages and adding artificial intelligence to the application as a project; In the third stage, it was planned to examine the effect of the application on the variables and scales. The data of the study were collected between June 2022 and June 2023 in the Endocrinology Polyclinic of two private hospitals in Izmir and a diabetes association where individuals with diabetes were registered. Power 0.80 was determined by using NCSS PAS statistical software from the population of the research; The minimum number of samples to be included in the study was calculated as n:122 and they were divided into two as intervention and control groups by randomization. The research sample was carried out as intervention (n:60) and control (n:60) lastly due to death and cost. Five data collection tools were used, namely "Individual Introduction Form", "Diabetes Self-Care Scale", "Hypoglycemia Confidence Scale", "Mobile Application Opinion Form" and "Cost Table". An artificial intelligence-based mobile virtual assistant application was applied to the individuals with diabetes in the intervention group, and the data were collected three times, at the 0th, 6th and 12th months, and the costs were recorded. The standard outpatient trainings, which are currently applied, continued to be given to individuals with diabetes in the control group, the data were collected twice, at the beginning (0. month) and 12. months, and the costs were recorded. In the evaluation of the data, number, percentage, arithmetic mean, standard deviation, minimum and maximum median were calculated. Among the variables, chi-square, Kruskal Wallis, Mann Whitney U test and t test were used.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 1 and Type 2 diabetes at least six months ago, according to the criteria of the American Diabetes Association (ADA),
* Using insulin for at least six months,
* Being between the ages of 18- 65,
* Being able to read and write and speak Turkish,
* Having an Android phone and being able to use mobile applications,
* To volunteer to participate in the study.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * The patient has a perception disorder and psychiatric disorder that prevents communication,
  * Desire to leave the research,
  * His death during the research,
  * Being pregnant,
  * Individuals with severe retinopathy and neuropathy that prevent smartphone use were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Care Scale | 12 months
  The score consists of 35 items and is a 4-point Likert type, the lowest acceptable score is 92 and the highest score is 140. As the score increases, self-care increases
Hypoglycemic Confidence Scale | 12 months
  The scale consists of 9 items and is a 4-point Likert type. There is no cut-off value, the average score is used.

SECONDARY OUTCOMES:
hospitalization rate | 12 months
  percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No